CLINICAL TRIAL: NCT00438464
Title: A Randomized Controlled Trial Evaluating the Tissue Effects of Preoperative Finasteride Versus Placebo for Patients With Clinically Organ-Confined Prostate Cancer
Brief Title: Finasteride in Treating Patients With Stage II Prostate Cancer Who Are Undergoing Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCI-2009-00856; NCI-2009-00856 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000653463; 2006-0614 (Other: M D Anderson Cancer Center); MDA03-1-03 (Other: DCP); N01CN35159 (NIH); P30CA016672 (NIH)
Record Dates: First submitted 2007-02-20; First posted 2007-02-22 (Estimated); Results first posted 2016-03-09 (Estimated); Last update posted 2016-03-09 (Estimated); Status verified 2015-06

CONDITIONS: Adenocarcinoma of the Prostate; Stage II Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Finasteride; Prostatectomy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (Finasteride) (Experimental): Finasteride 5 mg once daily for 4-6 weeks, then undergo prostatectomy.
  Interventions: Drug: Finasteride; Procedure: Prostatectomy; Other: Laboratory biomarker analysis
- Arm II (Placebo) (Placebo Comparator): Placebo once daily for 4-6 weeks, then undergo prostatectomy.
  Interventions: Other: Placebo; Other: Laboratory biomarker analysis

INTERVENTIONS:
Drug: Finasteride — Given PO
  Other Names: Finastid; MK 906; Proscar; Prostide
  Arms: Arm I (Finasteride)
Other: Placebo — Given PO
  Other Names: PLCB
  Arms: Arm II (Placebo)
Procedure: Prostatectomy — Undergo prostatectomy
  Other Names: Radical Prostatectomy; Therapeutic conventional surgery; Simple Prostatectomy
  Arms: Arm I (Finasteride)
Other: Laboratory biomarker analysis — Correlative studies

SUMMARY:
This randomized phase II trial studies how well finasteride works in treating patients with stage II prostate cancer who are undergoing surgery. Testosterone can cause the growth of prostate cancer cells. Hormone therapy using finasteride may fight prostate cancer by lowering the amount of testosterone the body makes. Giving finasteride before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Compare the frequency of discriminating molecular marker expression in Gleason grade (GG) 3 cores, adjusted for Gleason score (GS) at prostatectomy, in patients with stage II prostate cancer treated with neoadjuvant finasteride vs placebo.

SECONDARY OBJECTIVES:

I. Compare the frequency with which grade 3 and grade 4 tumors occur in these patients.

II. Determine the frequency of discriminating molecular signature expression in tissue microarray cores segregated by GS at prostatectomy in these patients.

III. Compare GG 3-appearing areas (in tumors rated GS 6 at prostatectomy) in patients treated with finasteride vs placebo.

IV. Compare GG 3-appearing areas (in tumors rated GS 7 at prostatectomy) in patients treated with finasteride vs placebo.

V. Compare GG 4-appearing areas (in tumors rated GS 7 at prostatectomy) in patients treated with finasteride vs placebo.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study.

Patients are stratified according to study site, Gleason score (6 vs 7), and type of prostatectomy (open vs robotic/laparoscopic). Patients are randomized to 1 of 2 treatment arms.

Arm I: Patients receive finasteride orally (PO) once daily (QD) for 4-6 weeks, and then undergo prostatectomy.

Arm II: Patients receive placebo PO QD for 4-6 weeks, and then undergo prostatectomy.

Tumor tissue obtained at prostatectomy is used to make tissue microarrays and is analyzed by immunohistochemistry for molecular marker expression studies.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Criteria:

* Histologically confirmed adenocarcinoma of the prostate
* Clinical stage T1c or T2 (stage II)
* Gleason score of 6 or 7 on initial biopsy
* Prostate-specific antigen (PSA) level less than 10 ng/mL within the past 3 months
* Candidate for and scheduled to undergo prostatectomy
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-2 OR Karnofsky PS 70-100%
* Fertile patients must use effective contraception
* No active malignancy at any other site
* No history of allergic reactions attributed to compounds of similar chemical or biological composition to finasteride
* No uncontrolled intercurrent illness including, but not limited to, any of the following: Ongoing or active infection; Symptomatic congestive heart failure; Unstable angina pectoris; Cardiac arrhythmia
* No psychiatric illness or social situation that would preclude study compliance
* More than 6 months since prior hormonal agents, including dutasteride or finasteride
* More than 6 months since prior chemotherapy
* More than 1 month since prior participation in another investigational study
* No prior radiotherapy for the primary tumor
* No concurrent dehydroepiandrosterone, phytoestrogen supplements, antiandrogen therapy, dutasteride, or other finasteride
* No concurrent anticoagulation, except for the use of daily acetylsalicylic acid (81 mg to 325 mg)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2007-02; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeri Kim, Principal Investigator — M.D. Anderson Cancer Center
Locations (8):
- United States (8):
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Audie L Murphy Veterans Affairs Hospital, San Antonio, Texas
  - Cancer Therapy and Research Center, San Antonio, Texas
  - University Hospital, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: From 2007 to 2012 recruitment was done at various medical clinic locations.
Pre-assignment Details: Of the 210 participants recruited, 204 were randomized to the study.
Period: Overall Study
Arm/Group | Arm I (Finasteride) | Arm II (Placebo)
Started | 103 | 101
Received Assigned Intervention | 89 | 94
Completed | 89 | 94
Not Completed | 14 | 7
Not completed — Terminated Early | 14 | 5
Not completed — Incomplete data submission | 0 | 2

BASELINE CHARACTERISTICS:
Population: Baseline includes participants who were randomized to arms and received assigned treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Finasteride) | Arm II (Placebo) | Total
Number analyzed (Participants) | 89 | 94 | 183
Age, Continuous [Median (Full Range); unit: years] | 59 [45 to 73] | 62 [48 to 73] | 60 [45 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 89 | 94 | 183
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 1 | 0 | 1
  Black | 5 | 7 | 12
  Hispanic | 5 | 2 | 7
  White | 78 | 85 | 163
Region of Enrollment [Number; unit: participants]
  United States | 89 | 94 | 183

OUTCOME MEASURES:

1. Secondary Outcome: Pathologic Characteristics of Radical Prostatectomy Specimens After Treatment: Gleason Score
Description: Frequency of Grade 3 and Grade 4 tumors in two treatment groups: Participants consist of men with adenocarcinoma of prostate, clinical stage T1c or T2, with Gleason score of 6 or 7 and PSA level < 10 ng/mL, who are scheduled to undergo prostatectomy. 2005 International Society of Urological Pathologists recommendations for Gleason scoring (GS) used to grade tumors based upon its microscopic appearance: a primary grade is assigned to most common tumor pattern, and a second grade to next most common tumor pattern. Gleason score (GS) is sum of the two Gleason grades, based on scale of 2-10 with lowest numbers indicating slow-growing tumor unlikely to spread and highest numbers indicating an aggressive tumor. Gleason grade = 1-5; Gleason score = 2-10; 5 and 10 indicate worst prognosis. American Joint Committee on Cancer (AJCC) staging describes extent of disease progression utilizing TNM scoring system: Tumor size, Lymph Nodes affected, Metastases. Higher stage cancers are more advanced.
Time Frame: Assessment following maximum 6 week treatment period and prostatectomy
Population: Analysis includes all evaluable participants. One participant in each arm was excluded due to hormonal therapy effect resulting in lack of assignment of Gleason Grade.
Measure: Number; unit: participants
Arm/Group | Arm I (Finasteride) | Arm II (Placebo)
Number analyzed (Participants) | 88 | 93
participants
  Gleason Score 6 | 12 | 10
  Gleason Score 7 | 71 | 78
  Gleason Score 8 | 2 | 1
  Gleason Score 9 | 3 | 4

2. Secondary Outcome: Pathologic Characteristics of Radical Prostatectomy Specimens After Treatment: Gleason Grade -- Specimen (Primary)
Description: Frequency of Grade 3 and Grade 4 tumors in two treatment groups: Participants consist of men with adenocarcinoma of the prostate, clinical stage T1c or T2, with a Gleason score of 6 or 7 and a PSA level < 10 ng/mL, who are scheduled to undergo prostatectomy.
Time Frame: Assessment following maximum 6 week treatment period and prostatectomy
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Arm I (Finasteride) | Arm II (Placebo)
Number analyzed (Participants) | 88 | 93
participants
  Grade 3 | 65 | 75
  Grade 4 | 23 | 18

3. Secondary Outcome: Pathologic Characteristics of Radical Prostatectomy Specimens After Treatment: Gleason Grade -- Specimen (Secondary)
Description: Frequency of Grade 3, Grade 4 and Grade 5 tumors in two treatment groups: Participants will consist of men with adenocarcinoma of the prostate, clinical stage T1c or T2, with a Gleason score of 6 or 7 and a PSA level < 10 ng/mL, who are scheduled to undergo prostatectomy.
Time Frame: Assessment following maximum 6 week treatment period and prostatectomy
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Arm I (Finasteride) | Arm II (Placebo)
Number analyzed (Participants) | 88 | 93
participants
  Grade 3 | 31 | 24
  Grade 4 | 53 | 64
  Grade 5 | 4 | 5

4. Secondary Outcome: Pathologic Characteristics of Radical Prostatectomy Specimens After Treatment: Tumor, Node, Metastasis (TNM) Stage
Description: American Joint Committee on Cancer (AJCC) system 6th edition (2002) describing amount and spread of cancer body, using TNM. T describes the size of the tumor and any spread of cancer into nearby tissue; N describes spread of cancer to nearby lymph nodes; and M describes metastasis (spread of cancer to other parts of the body). Numbers after the T (such as T1, T2, T3, and T4) describe tumor size and/or amount of spread into nearby structures. The higher the T number, the larger the tumor and/or the more it has grown into nearby tissues where T3a reflects tumor has spread through the capsule on one or both sides; and T3b reflects tumor has invaded one or both seminal vesicles.
Time Frame: Assessment following maximum 6 week treatment period and prostatectomy
Population: All evaluable participants.
Measure: Number; unit: participants
Arm/Group | Arm I (Finasteride) | Arm II (Placebo)
Number analyzed (Participants) | 89 | 94
participants
  pT2 | 73 | 74
  pT3a | 11 | 15
  pT3b | 5 | 5

5. Secondary Outcome: Pathologic Characteristics of Radical Prostatectomy Specimens After Treatment: Margin of Resection (MOR)
Description: Edge or border of tissue removed in cancer surgery. The margin is described as negative or clean when the pathologist finds no cancer cells at the edge of the tissue, suggesting that all of the cancer has been removed. The margin is described as positive or involved when the pathologist finds cancer cells at the edge of the tissue, suggesting that all of the cancer has not been removed.
Time Frame: Assessment following maximum 6 week treatment period and prostatectomy
Population: Analysis includes all evaluable participants.
Measure: Number; unit: participants
Arm/Group | Arm I (Finasteride) | Arm II (Placebo)
Number analyzed (Participants) | 89 | 94
participants
  Positive | 17 | 16
  Negative | 67 | 76
  Equivocal | 5 | 2

6. Secondary Outcome: Pathologic Characteristics of Radical Prostatectomy Specimens After Treatment: Lymph Node Status
Description: Status of cancer spread to lymph nodes; PN0 Cancer that has not spread to the lymph nodes. Cancer that has not spread to the lymph nodes. The N category describes whether the cancer has spread into nearby lymph nodes. NX means the nearby lymph nodes cannot be evaluated. N0 means nearby lymph nodes do not contain cancer. Numbers after the N (such as N1, N2, and N3) describe the size, location, and/or the number of nearby lymph nodes affected by cancer. The higher the N number, the greater the cancer spread to nearby lymph nodes.
Time Frame: Assessment following maximum 6 week treatment period and prostatectomy
Population: Analysis includes all evaluable participants.
Measure: Number; unit: participants
Arm/Group | Arm I (Finasteride) | Arm II (Placebo)
Number analyzed (Participants) | 89 | 94
participants
  PN0 | 46 | 43
  PN1 | 2 | 2
  pNX | 41 | 49

7. Secondary Outcome: Pathologic Characteristics of Radical Prostatectomy Specimens After Treatment: Cancer Foci
Description: Diagnosis of a small focus of prostatic adenocarcinoma on a prostate needle biopsy from pathologist's identification of an architecturally abnormal focus of epithelial structures at rather low magnification.
Time Frame: Assessment following maximum 6 week treatment period and prostatectomy
Population: Analysis includes all evaluable participants.
Measure: Number; unit: participants
Arm/Group | Arm I (Finasteride) | Arm II (Placebo)
Number analyzed (Participants) | 89 | 94
participants
  1 Focus | 15 | 11
  2 Foci | 18 | 20
  3 Foci | 28 | 28
  4 Foci | 13 | 20
  >/= 5 Foci | 15 | 15

8. Secondary Outcome: Pathologic Characteristics of Radical Prostatectomy Specimens After Treatment: Zonal Origin of Tumor Foci Per Radical Prostatectomy Specimen (RPS)
Description: Tumor distribution within zones of the prostate using radical prostatectomy specimen (RPS) where number of foci categorized by zone defined as: PZ, peripheral zone; TZ, transition zone; CZ, central zone.
Time Frame: Assessment following maximum 6 week treatment period and prostatectomy
Population: Analysis includes all evaluable participants.
Measure: Number; unit: participants
Arm/Group | Arm I (Finasteride) | Arm II (Placebo)
Number analyzed (Participants) | 89 | 94
participants
  PZ | 35 | 38
  PZ + TZ | 49 | 50
  PZ + TZ + CZ | 2 | 2
  PZ + CZ | 0 | 1
  TZ | 3 | 3

9. Secondary Outcome: Pathologic Characteristics of Radical Prostatectomy Specimens After Treatment: Zonal Origin -- Dominant Tumor Focus
Description: Dominant tumor focus, distribution within zones of the prostate using radical prostatectomy specimen (RPS) where number of foci categorized by zone defined as: PZ, peripheral zone; TZ, transition zone; CZ, central zone. Dominant tumor focus is the largest, index lesion, single high risk focus of the prostate cancer.
Time Frame: Assessment following maximum 6 week treatment period and prostatectomy
Population: Analysis includes all evaluable participants.
Measure: Number; unit: participants
Arm/Group | Arm I (Finasteride) | Arm II (Placebo)
Number analyzed (Participants) | 89 | 94
participants
  PZ | 67 | 73
  TZ | 22 | 21

10. Secondary Outcome: Pathologic Characteristics of Radical Prostatectomy Specimens After Treatment: Gleason Upgrade Between Biopsy and Prostatectomy
Description: Change in Gleason Score from biopsy to prostatectomy where an upgrade refers to a higher Gleason Score signifying worsening of tumor. Gleason scoring (GS) to based on microscopic appearance using 2005 International Society of Urological Pathologists recommendation.
Time Frame: Baseline biopsy to prostatectomy following maximum 6 week treatment period
Population: Analysis includes all evaluable participants.
Measure: Number; unit: participants
Arm/Group | Arm I (Finasteride) | Arm II (Placebo)
Number analyzed (Participants) | 89 | 94
participants
  No | 63 | 70
  Yes | 26 | 24

11. Secondary Outcome: Pathologic Characteristics of Radical Prostatectomy Specimens After Treatment: Tumor Volume (Cubic Centimeter)
Description: Characteristics of tumor considering total zone cancer volume, and cancer volume using zonal foci categorized as: PZ, peripheral zone; TZ, transition zone; CZ, central zone.
Time Frame: Baseline biopsy to prostatectomy following maximum 6 week treatment period
Population: Analysis includes all evaluable participants.
Measure: Median (Full Range); unit: cubic centimeter
Arm/Group | Arm I (Finasteride) | Arm II (Placebo)
Number analyzed (Participants) | 89 | 94
cubic centimeter
  Total | 1.0 [0.0 to 9.3] | 0.8 [0.0 to 10.4]
  PZ Cancer focus/foci | 0.6 [0.0 to 9.3] | 0.5 [0.0 to 9.0]
  TZ cancer focus/foci | 0.0 [0.0 to 6.0] | 0.0 [0.0 to 10.4]

12. Secondary Outcome: Characteristics of Blood Biomarkers: Prostate-specific Antigen (ng/mL) Percentage Change (%)
Description: Characteristics of blood biomarkers using pretreatment and posttreatment values. Prostate-specific antigen (PSA) blood test measuring protein produced by prostate cells.
Time Frame: Baseline biopsy to prostatectomy following maximum 6 week treatment period
Population: Analysis includes all evaluable participants.
Measure: Median (Full Range); unit: percentage of change
Arm/Group | Arm I (Finasteride) | Arm II (Placebo)
Number analyzed (Participants) | 75 | 80
percentage of change | -39.4 [-96.6 to 155.2] | -4.6 [-61.2 to 200.0]
Statistical Analysis 1: Comparison: Arm I (Finasteride) vs Arm II (Placebo); Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

13. Secondary Outcome: Characteristics of Blood Biomarkers: Testosterone (ng/dL) Percentage Change
Description: Characteristics of blood biomarkers using pretreatment and posttreatment values. Blood tests used for measuring the amount of testosterone in the blood.
Time Frame: Baseline biopsy to prostatectomy following maximum 6 week treatment period
Population: Analysis includes all evaluable participants.
Measure: Median (Full Range); unit: percentage of change
Arm/Group | Arm I (Finasteride) | Arm II (Placebo)
Number analyzed (Participants) | 76 | 80
percentage of change | 13 [-53 to 158] | -4.6 [-80.7 to 76.1]
Statistical Analysis 1: Comparison: Arm I (Finasteride) vs Arm II (Placebo); Test type: Superiority or Other; p = 0.003, Wilcoxon (Mann-Whitney)

14. Secondary Outcome: Characteristics of Blood Biomarkers: Dihydrotestosterone (ng/dL) Percentage Change
Description: Characteristics of blood biomarkers using pretreatment and posttreatment values. Dihydrotestosterone (DHT) blood test measures serum concentrations of dihydrotestosterone and is closely related to those of testosterone.
Time Frame: Baseline biopsy to prostatectomy following maximum 6 week treatment period
Population: Analysis includes all evaluable participants.
Measure: Median (Full Range); unit: percentage of change
Arm/Group | Arm I (Finasteride) | Arm II (Placebo)
Number analyzed (Participants) | 74 | 79
percentage of change | -64.8 [-90 to 120] | -3.6 [-64.7 to 615.1]
Statistical Analysis 1: Comparison: Arm I (Finasteride) vs Arm II (Placebo); Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

15. Secondary Outcome: Characteristics of Blood Biomarkers: Estrone (ng/dL) Percentage Change
Description: Characteristics of blood biomarkers using pretreatment and posttreatment values. Blood test used to measure Estrone (E1), one of the three estrogens, which also includes estriol and estradiol.
Time Frame: Baseline biopsy to prostatectomy following maximum 6 week treatment period
Population: Analysis includes all evaluable participants.
Measure: Median (Full Range); unit: percentage of change
Arm/Group | Arm I (Finasteride) | Arm II (Placebo)
Number analyzed (Participants) | 75 | 79
percentage of change | -8.9 [-93.2 to 870] | 0 [-81.8 to 760]
Statistical Analysis 1: Comparison: Arm I (Finasteride) vs Arm II (Placebo); Test type: Superiority or Other; p = 0.805, Wilcoxon (Mann-Whitney)

16. Secondary Outcome: Characteristics of Blood Biomarkers: Estradiol (ng/dL) Percentage Change
Description: Characteristics of blood biomarkers using pretreatment and posttreatment values. Blood test used to measure Estradiol.
Time Frame: Baseline biopsy to prostatectomy following maximum 6 week treatment period
Population: Analysis includes all evaluable participants.
Measure: Median (Full Range); unit: percentage of change
Arm/Group | Arm I (Finasteride) | Arm II (Placebo)
Number analyzed (Participants) | 76 | 79
percentage of change | 7.2 [-80.0 to 700] | 0 [-86.8 to 161.5]
Statistical Analysis 1: Comparison: Arm I (Finasteride) vs Arm II (Placebo); Test type: Superiority or Other; p = 0.254, Wilcoxon (Mann-Whitney)

17. Primary Outcome: Comparison of Biomarkers Between Treatment Arms: Percentage Change of Tumor Cells Exhibiting Detectable Staining Within Gleason Grade 3 (GG3) Biomarker Subgroups at Prostatectomy
Description: Molecular marker expression based on tissue microarray (TMA) derived from dominant tumor focus. Staining microarrays for high-throughput assessment of candidate gene expression and data modeling constructed with a tissue microarray apparatus and 0.6-mm biopsy cores, representative of tumor grades and scores (Gleason Grades 3 (GG3) and Gleason Grade 4 (GG4)). The percentage of tumor cells exhibiting detectable staining, scored as 0 to 10 where higher score designates more involvement, as applicable for: vascular epithelial growth factor (VEFG), estrogen receptor beta (ERβ), androgen receptor (AR), 3-oxo-5α-steroid 4-dehydrogenase 2 (SRD5A2), ubiquitin-conjugating enzyme E2C (UBE2C), and Cleaved Caspase 3 (Caspase). P values are based on non-parametric Wilcoxon rank-sum test.
Time Frame: At prostatectomy following maximum 6 week treatment period
Population: Of total 183 enrolled participants in both arms, 62 Finasteride and 68 Placebo participants respectively had a qualifying tumor specimen with GG3 or GG4. Differences in number (N) of tissue specimens (tumor foci) is based on feasibility of subgroup participants' radical prostatectomy samples analyzed.
Measure: Median (Full Range); unit: Percentage tumor cell involvement
Groups:
- Finasteride Arm Within GG3: Finasteride 5 mg once daily for 4-6 weeks, then undergo prostatectomy.
- Placebo Arm Within GG3: Placebo once daily for 4-6 weeks, then undergo prostatectomy.
Arm/Group | Finasteride Arm Within GG3 | Placebo Arm Within GG3
Number analyzed (Participants) | 62 | 68
Percentage tumor cell involvement
  VEGF (N=37,55) | 80 [5 to 100] | 90 [0 to 100]
  ERβ (N=35, 55) | 15.0 [0.03 to 59.0] | 6.6 [0 to 56.3]
  AR (N=35, 54) | 75.2 [21.5 to 92.1] | 78.3 [33.8 to 97.6]
  Ki-67 (N=37,54) | 1.1 [0.05 to 5.4] | 1.3 [0.03 to 4.5]
  SRD5A2 (N=45,47) | 100 [0 to 100] | 90 [0 to 100]
  UBE2C (N=34,55) | 0.4 [0 to 1.5] | 0.3 [0 to 2.4]
  Caspase (N=38,55) | 0.2 [0.01 to 4.1] | 0.08 [0 to 0.8]
Statistical Analysis 1: Comparison: Finasteride Arm Within GG3 vs Placebo Arm Within GG3; VEGF3, Within GG3; Test type: Superiority or Other; p = 0.70, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Finasteride Arm Within GG3 vs Placebo Arm Within GG3; Estrogen receptor beta (ERβ), Within GG3; Test type: Superiority or Other; p = 0.38, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Finasteride Arm Within GG3 vs Placebo Arm Within GG3; Androgen receptor (AR), Within GG3; Test type: Superiority or Other; p = 0.41, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Finasteride Arm Within GG3 vs Placebo Arm Within GG3; Ki-67 protein, Within GG3; Test type: Superiority or Other; p = 0.75, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Finasteride Arm Within GG3 vs Placebo Arm Within GG3; 3-oxo-5α-steroid 4-dehydrogenase 2 (SRD5A2), Within GG3; Test type: Superiority or Other; p = 0.57, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Finasteride Arm Within GG3 vs Placebo Arm Within GG3; Ubiquitin-conjugating enzyme E2C (UBE2C), Within GG3; Test type: Superiority or Other; p = 0.12, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Finasteride Arm Within GG3 vs Placebo Arm Within GG3; Cleaved Caspase 3 (Caspase), Within GG3; Test type: Superiority or Other; p = 0.03, Wilcoxon (Mann-Whitney)

18. Primary Outcome: Comparison of Biomarkers Between Treatment Arms: Percentage Change of Tumor Cells Exhibiting Detectable Staining Within Gleason Grade 4 (GG4) Biomarker Subgroup at Prostatectomy
Description: Biomarkers using pretreatment and posttreatment values. Staining microarrays for high-throughput assessment of candidate gene expression and data modeling constructed with a tissue microarray apparatus and 0.6-mm biopsy cores, representative of tumor grades and scores (Gleason Grades 3 (GG3) and Gleason Grade 4 (GG4)). The percentage of tumor cells exhibiting detectable staining, scored as 0 to 10 where higher score designates more involvement, as applicable for: VEGF denotes vascular epithelial growth factor, ERβ estrogen receptor beta, AR androgen receptor, SRD5A2, 3-oxo-5α-steroid 4-dehydrogenase 2, UBE2C, ubiquitin-conjugating enzyme E2C. P values are based on non-parametric Wilcoxon rank-sum test.
Time Frame: At prostatectomy following maximum 6 week treatment period
Population: as for outcome 17
Measure: Median (Full Range); unit: Percentage of tumor cell involvement
Groups:
- Finasteride Arm Within GG4: Finasteride 5 mg once daily for 4-6 weeks, then undergo prostatectomy.
- Placebo Arm Within GG4: Placebo once daily for 4-6 weeks, then undergo prostatectomy.
Arm/Group | Finasteride Arm Within GG4 | Placebo Arm Within GG4
Number analyzed (Participants) | 62 | 68
Percentage of tumor cell involvement
  VEGF (N=48,61) | 85 [5 to 100] | 70 [0 to 100]
  ERβ (N=48,62) | 8.0 [0 to 49.6] | 9.5 [0 to 72.8]
  AR (N=48,62) | 63.71 [13.5 to 92.0] | 75.9 [1.4 to 96.6]
  Ki-67 (N=48,62) | 1.3 [0.05 to 7.2] | 1.4 [0.05 to 7.3]
  SRD5A2 (N=38,69) | 95 [0 to 100] | 90 [0 to 100]
  UBE2C (N=46,62) | 0.3 [0 to 1.6] | 0.3 [0 to 2.3]
  Caspase (N=47,61) | 0.06 [0 to 0.5] | 0.04 [0 to 0.6]
Statistical Analysis 1: Comparison: Finasteride Arm Within GG4 vs Placebo Arm Within GG4; Vascular Epithelial Growth Factor (VEGF3), Within GG4; Test type: Superiority or Other; p = 0.45, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Finasteride Arm Within GG4 vs Placebo Arm Within GG4; Estrogen receptor beta (ERβ), Within GG4; Test type: Superiority or Other; p = 0.83, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Finasteride Arm Within GG4 vs Placebo Arm Within GG4; Androgen receptor (AR), Within GG4; Test type: Superiority or Other; p = 0.04, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Finasteride Arm Within GG4 vs Placebo Arm Within GG4; Ki-67 protein, Within GG4; Test type: Superiority or Other; p = 0.80, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Finasteride Arm Within GG4 vs Placebo Arm Within GG4; 3-oxo-5α-steroid 4-dehydrogenase 2 (SRD5A2), Within GG4; Test type: Superiority or Other; p = 0.61, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Finasteride Arm Within GG4 vs Placebo Arm Within GG4; UBE2C, Within GG4; Test type: Superiority or Other; p = 0.86, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Finasteride Arm Within GG4 vs Placebo Arm Within GG4; Caspase, Within GG4; Test type: Superiority or Other; p = 0.02, Wilcoxon (Mann-Whitney)

19. Primary Outcome: Comparison of Biomarkers Between Treatment Arms: Percentage Change of Tumor Cells Exhibiting Detectable Staining Within Gleason Grade 3 (GG3) Biomarker Subgroups at Prostatectomy
Description: Molecular marker expression compared between tumor foci using Biomarkers pretreatment and posttreatment values. Staining microarrays for high-throughput assessment of candidate gene expression and data modeling constructed with a tissue microarray apparatus and 0.6-mm biopsy cores, representative of tumor grades and scores (Gleason Grades 3 (GG3) and Gleason Grade 4 (GG4)). The percentage of tumor cells exhibiting detectable staining, scored as 0 to 10 where higher score designates more involvement, as applicable for: VEGF denotes vascular epithelial growth factor, ERβ estrogen receptor beta, AR androgen receptor, SRD5A2, 3-oxo-5α-steroid 4-dehydrogenase 2, UBE2C, ubiquitin-conjugating enzyme E2C.
Time Frame: At prostatectomy following maximum 6 week treatment period.
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Percentage of tumor cell involvement
Arm/Group | Finasteride Arm Within GG3 | Placebo Arm Within GG3
Number analyzed (Participants) | 62 | 68
Percentage of tumor cell involvement
  VEGF (N=37,55) | 63.9 (36.3) | 63.7 (38)
  ERβ (N=35, 55) | 18.1 (15.6) | 14.8 (14.7)
  AR (N=35, 54) | 69.8 (17.3) | 72.4 (16.7)
  Ki-67 (N=37,54) | 1.6 (1.4) | 1.5 (1.0)
  SRD5A2 (N=45,47) | 72.9 (37.0) | 64.7 (43.7)
  UBE2C (N=34,55) | 0.5 (0.4) | 0.5 (0.5)
  Caspase (N=38,55) | 0.4 (0.7) | 0.2 (0.2)

20. Primary Outcome: Comparison of Biomarkers Between Treatment Arms: Percentage Change of Tumor Cells Exhibiting Detectable Staining Within Gleason Grade 4 (GG4) Biomarker Subgroup at Prostatectomy
Description: as for outcome 19
Time Frame: At prostatectomy following maximum 6 week treatment period.
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Percentage of tumor cell involvement
Arm/Group | Finasteride Arm Within GG4 | Placebo Arm Within GG4
Number analyzed (Participants) | 62 | 68
Percentage of tumor cell involvement
  VEGF (N=48,61) | 63.6 (35.5) | 59.8 (35.4)
  ERβ (N=48,62) | 15.0 (15.1) | 16.7 (18.8)
  AR (N=48,62) | 64.3 (16.67) | 68.6 (23.1)
  Ki-67 (N=48,62) | 1.8 (1.6) | 1.7 (1.4)
  SRD5A2 (N=38,69) | 71.8 (37.6) | 64.9 (40.8)
  UBE2C (N=46,62) | 0.5 (0.4) | 0.5 (0.4)
  Caspase (N=47,61) | 0.1 (0.1) | 0.06 (0.08)

21. Secondary Outcome: Comparison of Biomarkers Between Gleason Grades GG3 & GG4: Percentage of Tumor Cells Exhibiting Detectable Staining Within Finasteride Treatment Arm for Biomarker Subgroups (Mean)
Description: Molecular marker expression compared between tumor foci, characteristics of blood biomarkers using pretreatment and posttreatment values. VEGF denotes vascular epithelial growth factor, ERβ estrogen receptor beta, AR androgen receptor, SRD5A2, 3-oxo-5α-steroid 4-dehydrogenase 2, UBE2C, ubiquitin-conjugating enzyme E2C.
Time Frame: At prostatectomy following maximum 6 week treatment period
Population: Of total 89 enrolled participants in the Finasteride Arm, 62 participants had either a qualifying tumor specimen with GG3 or GG4. Differences in number (N) of tissue specimens (tumor foci) is based on feasibility of subgroup participants' radical prostatectomy samples analyzed.
Measure: Mean (Standard Deviation); unit: Percentage of tumor cell involvement
Groups:
- GG3, Within Finasteride Arm: Participants with GG3 score receiving 5 mg daily for 4-6 weeks, then receive prostatectomy.
- GG4, Within Finasteride Arm: Participants with GG4 score receiving 5 mg daily for 4-6 weeks, then receive prostatectomy.
Arm/Group | GG3, Within Finasteride Arm | GG4, Within Finasteride Arm
Number analyzed (Participants) | 62 | 62
Percentage of tumor cell involvement
  VEGF (N=37,48) | 63.9 (36.3) | 63.7 (35.5)
  ERβ (N=35,48) | 18.1 (15.6) | 15.0 (15.1)
  AR (N=35,48) | 69.8 (17.3) | 64.3 (16.7)
  Ki-67 (N=37,48) | 1.6 (1.4) | 1.8 (1.6)
  SRD5A2 (N=45,38) | 72.9 (37.0) | 71.8 (37.6)
  UBE2C (N=34,46) | 0.5 (0.4) | 0.5 (0.4)
  Caspase (N=38,47) | 0.4 (0.7) | 0.1 (0.1)

22. Secondary Outcome: Comparison of Biomarkers Between Gleason Grades GG3 & GG4: Percentage of Tumor Cells Exhibiting Detectable Staining Within Placebo Treatment Arm for Biomarker Subgroups (Mean)
Description: as for outcome 21
Time Frame: At prostatectomy following maximum 6 week treatment period.
Population: Of total 94 enrolled participants in the Placebo Arm, 68 participants had either a qualifying tumor specimen with GG3 or GG4. Differences in number (N) of tissue specimens (tumor foci) is based on feasibility of subgroup participants' radical prostatectomy samples analyzed.
Measure: Mean (Standard Deviation); unit: Percentage of tumor cell involvement
Groups:
- GG3, Within Placebo Arm: Participants with GG3 score in Placebo Arm, receiving placebo daily for 4-6 weeks, then receive prostatectomy.
- GG4, Within Placebo Arm: Participants with GG4 score in Plaebo Arm, receiving placebo daily for 4-6 weeks, then receive prostatectomy.
Arm/Group | GG3, Within Placebo Arm | GG4, Within Placebo Arm
Number analyzed (Participants) | 68 | 68
Percentage of tumor cell involvement
  VEGF (N=55,61) | 63.7 (38) | 59.7 (35.4)
  ERβ (N=55,62) | 14.8 (14.7) | 16.7 (18.8)
  AR (N=54,62) | 72.4 (16.7) | 68.6 (23.1)
  Ki-67 (N=54,62) | 1.5 (1.0) | 1.7 (1.4)
  SRD5A2 (N=47,69) | 64.7 (43.7) | 64.9 (40.8)
  UBE2C (N=55,62) | 0.5 (0.5) | 0.5 (0.4)
  Caspase (N=55,61) | 0.2 (0.2) | 0.06 (0.08)

23. Secondary Outcome: Comparison of Biomarkers Between Gleason Grades GG3 & GG4: Percentage of Tumor Cells Exhibiting Detectable Staining Within Finasteride Treatment Arm for Biomarker Subgroups
Description: Molecular marker expression compared between tumor foci, characteristics of blood biomarkers using pretreatment and posttreatment values. VEGF denotes vascular epithelial growth factor, ERβ estrogen receptor beta, AR androgen receptor, SRD5A2, 3-oxo-5α-steroid 4-dehydrogenase 2, UBE2C, ubiquitin-conjugating enzyme E2C. P values are based on non-parametric Wilcoxon rank-sum test.
Time Frame: At prostatectomy following maximum 6 week treatment period
Population: as for outcome 21
Measure: Median (Full Range); unit: Percentage of tumor cell involvement
Groups:
- Within GG3, Finasteride Arm: Participants with GG3 score in Finasteride Arm, receiving 5 mg daily for 4-6 weeks, then receive prostatectomy.
- Within GG4, Finasteride Arm: Participants with GG4 score in Finasteride Arm, receiving 5 mg daily for 4-6 weeks, then receive prostatectomy.
Arm/Group | Within GG3, Finasteride Arm | Within GG4, Finasteride Arm
Number analyzed (Participants) | 62 | 62
Percentage of tumor cell involvement
  VEGF (N=37,48) | 80 [5 to 100] | 85 [5 to 100]
  ERβ (N=35,48) | 15.0 [0.03 to 58.9] | 8.0 [0 to 49.56]
  AR (N=35,48) | 75.2 [21.5 to 92.1] | 63.7 [13.5 to 92.0]
  Ki-67 (N=37,48) | 1.1 [0.05 to 5.4] | 1.3 [0.05 to 7.2]
  SRD5A2 (N=45,38) | 100 [0 to 100] | 95 [0 to 100]
  UBE2C (N=34,46) | 0.4 [0 to 1.5] | 0.3 [0 to 1.6]
  Caspase (N=38,47) | 0.2 [0.01 to 4.1] | 0.06 [0 to 0.5]
Statistical Analysis 1: Comparison: Within GG3, Finasteride Arm vs Within GG4, Finasteride Arm; VEGF3, Within Finasteride Arm; Test type: Superiority or Other; p = 0.84, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Within GG3, Finasteride Arm vs Within GG4, Finasteride Arm; ERβ, Within Finasteride Arm; Test type: Superiority or Other; p = 0.36, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Within GG3, Finasteride Arm vs Within GG4, Finasteride Arm; AR, Within Finasteride; Test type: Superiority or Other; p = 0.09, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Within GG3, Finasteride Arm vs Within GG4, Finasteride Arm; Ki-67 protein, Within Finasteride Arm; Test type: Superiority or Other; p = 0.46, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Within GG3, Finasteride Arm vs Within GG4, Finasteride Arm; SRD5A2, Within Finasteride Arm; Test type: Superiority or Other; p = 0.88, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Within GG3, Finasteride Arm vs Within GG4, Finasteride Arm; UBE2C, Within Finasteride Arm; Test type: Superiority or Other; p = 0.18, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Within GG3, Finasteride Arm vs Within GG4, Finasteride Arm; Caspase, Within Finasteride Arm; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

24. Secondary Outcome: Comparison of Biomarkers Between Gleason Grades GG3 & GG4: Percentage of Tumor Cells Within Placebo Treatment Arm for Biomarker Subgroups
Description: as for outcome 23
Time Frame: At prostatectomy following maximum 6 week treatment period.
Population: as for outcome 22
Measure: Median (Full Range); unit: Percentage of tumor cell involvement
Groups:
- Within GG3, Placebo Arm: Participants with GG3 score in Placebo Arm, receiving placebo daily for 4-6 weeks, then receive prostatectomy.
- Within GG4, Placebo Arm: Participants with GG4 score in Plaebo Arm, receiving placebo daily for 4-6 weeks, then receive prostatectomy.
Arm/Group | Within GG3, Placebo Arm | Within GG4, Placebo Arm
Number analyzed (Participants) | 68 | 68
Percentage of tumor cell involvement
  VEGF (N=55,61) | 90 [0 to 100] | 70 [0 to 100]
  ERβ (N=55,62) | 6.6 [0 to 56.3] | 9.5 [0 to 72.8]
  AR (N=54,62) | 78.3 [33.77 to 97.6] | 75.9 [1.39 to 96.6]
  Ki-67 (N=54,62) | 1.3 [0.03 to 4.5] | 1.4 [0.05 to 7.3]
  SRD5A2 (N=47,69) | 90 [0 to 100] | 90 [0 to 100]
  UBE2C (N=55,62) | 0.3 [0 to 2.4] | 0.3 [0 to 2.3]
  Caspase (N=55,61) | 0.08 [0 to 0.8] | 0.04 [0 to 0.6]
Statistical Analysis 1: Comparison: Within GG3, Placebo Arm vs Within GG4, Placebo Arm; VEGF3, Within Placebo Arm; Test type: Superiority or Other; p = 0.32, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Within GG3, Placebo Arm vs Within GG4, Placebo Arm; ERβ, Within Placebo Arm; Test type: Superiority or Other; p = 0.83, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Within GG3, Placebo Arm vs Within GG4, Placebo Arm; AR, Within Placebo Arm; Test type: Superiority or Other; p = 0.77, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Within GG3, Placebo Arm vs Within GG4, Placebo Arm; Ki-67 protein, Within Placebo Arm; Test type: Superiority or Other; p = 0.87, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Within GG3, Placebo Arm vs Within GG4, Placebo Arm; SRD5A2, Within Placebo Arm; Test type: Superiority or Other; p = 0.91, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Within GG3, Placebo Arm vs Within GG4, Placebo Arm; UBE2C, Within Placebo Arm; Test type: Superiority or Other; p = 0.90, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Within GG3, Placebo Arm vs Within GG4, Placebo Arm; Caspase, Within Placebo Arm; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: The final collection of adverse events obtained at the completion of the 4-6 week course of study medication/placebo, before prostatectomy. Overall study period: March 2007 to April 2012.
Arm/Group | Arm I (Finasteride) | Arm II (Placebo)
Serious Adverse Events (participants affected / at risk) | 0/89 | 0/94
Other Adverse Events (participants affected / at risk) | 0/89 | 0/94

LIMITATIONS AND CAVEATS:
Predefined molecular signature could not easily distinguish GG 4 from GG 3 tumor areas in the placebo arm.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less